CLINICAL TRIAL: NCT04346537
Title: INGEVITY+ Active Fixation Pace/Sense Lead Clinical Study
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 92424682
Record Dates: First submitted 2020-04-08; First posted 2020-04-15 (Actual); Results first posted 2022-05-12 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: INGEVITY+™ Pace/Sense Lead — The INGEVITY+ lead is indicated for chronic pacing and sensing in the right atrium and/or right ventricle when used with a compatible pulse generator.

SUMMARY:
The objective of this study is it to confirm the safety and effectiveness of the INGEVITY+ Active Fixation Pace/Sense Lead.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and capable of providing informed consent
2. Subject is intended to undergo initial (de novo) pacing system implant using INGEVITY+ Leads in the Right Atrium (RA) and Right Ventricle (RV) and a Boston Scientific pulse generator
3. Subject meets an indication for a Boston Scientific Pacemaker or CRT-P device per product labeling (Physician's Technical Manual)
4. Willing and capable of participating in all testing/visits associated with this clinical study at an approved clinical study center and at the intervals defined by this protocol
5. Age 18 or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

1. Known or suspected sensitivity to dexamethasone acetate (DXA)
2. Has a mechanical tricuspid heart valve
3. Women of childbearing potential who are or might be pregnant at the time of study enrollment or INGEVITY+ Lead implant (method of assessment upon physician's discretion)
4. Currently requiring hemo- or peritoneal dialysis
5. Subject has or has had implanted any pacing or ICD system, including subcutaneous, transvenous or leadless systems
6. Intended to receive a single chamber device
7. Documented history of permanent or persistent AF
8. Currently on an active organ transplant list
9. Documented life expectancy of less than 12 months
10. Enrolled in any other concurrent study unless prior approval is received from the Sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from the investigator's general patient population indicated for dual-chamber pacemaker or CRT-P implantation.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devi Nair, MD, Principal Investigator — Arrhythmia Research Group
Locations (13):
- United States (13):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Torrance Memorial Medical Center, Torrance, California
  - Emory University Hospital, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cardiovascular Institute of Michigan, Clinton Township, Michigan
  - Cox Health, Springfield, Missouri
  - Catholic Medical Center, Manchester, New Hampshire
  - Deborah Heart and Lung, Browns Mills, New Jersey
  - Aultman Hospital, Canton, Ohio
  - Saint Thomas Health, Nashville, Tennessee
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - PeaceHealth Southwest Medical, Bellingham, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Leads
Groups:
- INGEVITY+ Study Participants: Each participant was allowed to have up to 2 INGEVITY+ leads contribute to endpoint analyses -- one per chamber (right atrium and right ventricle). Final lead implanted or attempted during initial procedure per chamber was used for analysis.
Period: Overall Study
Arm/Group | INGEVITY+ Study Participants
Started | 109; 201 Leads (8 subjects did not undergo the implant procedure and did not have the INGEVITY+ lead implanted or attempted.)
Implanted/Attempted With INGEVITY+ Lead | 101; 201 Leads
Completed | 99; 198 Leads
Not Completed | 10; 3 Leads

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported on enrolled participants.
Groups:
- INGEVITY+ Study Participants: Enrolled INGEVITY+ Study Participants
Arm/Group | INGEVITY+ Study Participants
Number analyzed (Participants) | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 108
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 96
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 109
Brady Arrhythmia History [Count of Participants; unit: Participants]
  Sinus Bradycardia | 72
  Sinus Node Dysfunction | 29
  Chronotropic Incompetence | 7
  Sinus Arrest | 4
  Atrioventricular Block - 1st Degree | 4
  Atrioventricular Block - 2nd Degree (Intermittent) | 5
  Atrioventricular Block - 2nd Degree (Permanent) | 6
  Atrioventricular Block - 3rd Degree (Intermittent) | 2
  Atrioventricular Block - 3rd Degree (Permanent) | 4

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety: Lead-related Complication-Free Rate
Description: This endpoint evaluated the percentage of leads free from complication from three months post-implant through twelve months post implant. The performance goal was 93%. Kaplan-Meier methodology was used to calculate the complication-free rate %.
Time Frame: Lead Implant through 3-Months Post-Implant
Measure: Number (97.5% Confidence Interval); unit: Percentage of leads
Units Other Than Participants: Leads
Groups:
- INGEVITY+ Leads: Final lead implanted or attempted during initial procedure per chamber was used for analysis. Analysis leads were from participants who were implanted or attempted with INGEVITY+ lead(s). Of the 109 enrolled participants, there were 201 leads (101 implanted in right atrium, 99 implanted in right ventricle, 1 attempted in right ventricle) that met the eligibility criteria for inclusion in endpoint analyses.
Arm/Group | INGEVITY+ Leads
Number analyzed (Participants) | 101
Number analyzed (Leads) | 201
Percentage of leads | 98.5 [95.4 to NA] — Pre-specified analysis required lower one-sided confidence interval to be compared to performance goal of 93%. Upper confidence interval was irrelevant for endpoint analysis.

2. Primary Outcome: Primary Efficacy: Pacing Capture Threshold Responder Rate
Description: This endpoint evaluated the % of leads with an adequate INGEVITY+ Pacing Capture Threshold (PCT) measurement. A lead with an adequate INGEVITY+ PCT measurement was referred to as a Pacing Capture Threshold Responder. A responder was defined by a PCT at 3-month visit ≤ 2 V, measured at 0.4 ms pulse width. A performance goal of 80% was used.
Time Frame: At 3-Months Post-Implant
Population: Of the 201 leads eligible for endpoint analysis, 15 did not contribute to data the analysis (1 had unsuccessful lead implant, 14 had missing 3 month data due to death/withdrawal prior to 3-month visit, missed 3-month visit or incomplete lead measurement data).
Measure: Number (95% Confidence Interval); unit: Percentage of leads
Units Other Than Participants: Leads
Groups:
- INGEVITY+ Leads: Final lead implanted or attempted during initial procedure per chamber was used for analysis. Analysis leads were from participants who were implanted or attempted with INGEVITY+ lead(s). Of the 109 enrolled participants, there were 201 leads (101 implanted in right atrium, 99 implanted in right ventricle and 1 attempted in right ventricle) that met the eligibility criteria for inclusion in endpoint analyses.
Arm/Group | INGEVITY+ Leads
Number analyzed (Participants) | 98
Number analyzed (Leads) | 186
Percentage of leads | 98.9 [96.2 to 99.9]

3. Secondary Outcome: Secondary Efficacy: Sensed Amplitude in mV (Right Atrial Leads)
Description: This secondary endpoint evaluated the sensed amplitudes at 3-months post-implant. Atrial and ventricular leads were evaluated separately. The performance goal for atrial leads was > 1.5 mV.
Time Frame: At 3-Months Post-Implant
Population: Of the 101 right atrial leads eligible for endpoint analysis, 9 did not contribute to data the analysis due to death/withdrawal prior to 3-month visit, missed 3-month visit or incomplete lead measurement data.
Measure: Median (Inter-Quartile Range); unit: millivolts
Units Other Than Participants: Right Atrial Leads
Arm/Group | INGEVITY+ Leads
Number analyzed (Participants) | 92
Number analyzed (Right Atrial Leads) | 92
millivolts | 4.3 [2.4 to 6.2]
Statistical Analysis 1: Comparison: INGEVITY+ Leads; Test type: Superiority; p < 0.001, Wilcoxon signed rank test

4. Secondary Outcome: Secondary Efficacy: Sensed Amplitude in mV (Right Ventricular Leads)
Description: This secondary endpoint evaluated the sensed amplitudes at 3-months post-implant. Atrial and ventricular leads were evaluated separately. The performance goal for ventricular leads was > 1.5 mV.
Time Frame: At 3-Months Post-Implant
Population: Of the 100 right ventricular leads eligible for endpoint analysis, 12 did not contribute to data the analysis (1 had unsuccessful lead implant, 11 had missing 3 month data due to death/withdrawal prior to 3-month visit, missed 3-month visit or incomplete lead measurement data).
Measure: Median (Inter-Quartile Range); unit: millivolts
Units Other Than Participants: Right Ventricular Leads
Arm/Group | INGEVITY+ Leads
Number analyzed (Participants) | 88
Number analyzed (Right Ventricular Leads) | 88
millivolts | 15.9 [10.5 to 24.0]
Statistical Analysis 1: Comparison: INGEVITY+ Leads; Test type: Superiority; p < 0.001, Wilcoxon signed rank test

5. Secondary Outcome: Secondary Efficacy: Pacing Impedance in Ohms
Description: This secondary endpoint evaluated the pacing impedances at 3-months post-implant. The performance goals were > 300 ohms and < 1300 ohms.
Time Frame: At 3-Months Post-Implant
Population: Of the 201 leads eligible for endpoint analysis, 5 did not contribute to data the analysis (1 had unsuccessful lead implant, 4 had missing 3 month data due to death/withdrawal prior to 3-month visit, missed 3-month visit or incomplete lead measurement data).
Measure: Mean (90% Confidence Interval); unit: ohms
Units Other Than Participants: Leads
Arm/Group | INGEVITY+ Leads
Number analyzed (Participants) | 99
Number analyzed (Leads) | 196
ohms | 712 [696 to 729]
Statistical Analysis 1: Comparison: INGEVITY+ Leads; Test type: Other — Two-one sided t-tests (TOST) -- the 90% confidence interval was required to be contained with 300 and 1300 ohms; p < 0.001, Two one-sided t-tests

ADVERSE EVENTS:
Time Frame: Implant through 3-months post-implant.
Description: Only subjects implanted or attempted with an INGEVITY+ lead were considered at risk for an adverse event (N = 101).
Arm/Group | INGEVITY+ Study Participants
All-Cause Mortality (participants affected / at risk) | 1/101
Serious Adverse Events (participants affected / at risk) | 8/101
Other Adverse Events (participants affected / at risk) | 10/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INGEVITY+ Study Participants (N=101)
Dislodgment - related to right atrial lead (Product Issues) | 1 (1)
Myocardial perforation post-implant - related right atrial lead (Product Issues) | 1 (1)
Hemothorax (Surgical and medical procedures) | 1 (1)
Post-surgical infection (<=30 days post-implant) (Surgical and medical procedures) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Death (General disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Systemic infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INGEVITY+ Study Participants (N=101)
Sensation of pacing with auto threshold - related to pulse generator (Product Issues) | 1 (1)
Dislodgment - related to right atrial lead (Product Issues) | 1 (1)
Dislodgment - related to right ventricular lead (Product Issues) | 1 (2)
Adverse reaction (Surgical and medical procedures) | 2 (2)
Chest pain (Surgical and medical procedures) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrial tachycardia/Other supraventricular tachycardia (Cardiac disorders) | 1 (1)
Deep vein thrombosis (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction on the PI that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is equal to 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. Sponsor reserves the right to require deletion of any Confidential Information or other proprietary information of Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT04346537/Prot_SAP_000.pdf